CLINICAL TRIAL: NCT07089784
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Multiple Doses of MK-2828 in Participants With Type 2 Diabetes
Brief Title: Multiple Dose Study of MK-2828 in Participants With Type 2 Diabetes (MK-2828-003)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2828-003
Record Dates: First submitted 2025-07-25; First posted 2025-07-28 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MK-2828 (Experimental): Participants receive daily MK-2828 for 28 days.
  Interventions: Drug: MK-2828
- Placebo (Placebo Comparator): Participants receive daily placebo for 28 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-2828 — Oral capsule of MK-2828 taken once per day for 28 days.
  Arms: MK-2828
Drug: Placebo — Placebo to match MK-2828 oral capsule, taken once per day for 28 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to learn about the safety and if people tolerate a study medicine called MK-2828. The study will also measure what happens to MK-2828 in the body of a person with type 2 diabetes (T2D) over time (pharmacokinetic or PK study), and how it affects the amount of high-sensitivity C-reactive protein (hsCRP) in a person's blood.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* With the exception of type 2 diabetes mellitus (T2DM), is in generally good health
* Has a history of T2DM for ≥1 year at the time of screening based on self-reporting
* Has a baseline HbA1C level of ≤10% at the time of screening
* Has a stable weight (based on self-reporting) defined as ≤5 kg gain or loss of body weight for at least 3 months before Visit 1/Screening
* T2DM treated with lifestyle modification alone or with stable doses (no significant change for ≥3 months from Visit 1/Screening, based on self-reporting) of ≤ 3 oral anti-diabetic medications and anticipated not to require dose adjustments during the study duration
* Body mass index (BMI) between 25 and 40 kg/m2, inclusive

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has known systemic hypersensitivity to the MK-2828 drug substance or other nucleotide-binding, leucine-rich, protein 3 inhibitor (NLRP3i) based therapy, its inactive ingredients, or the placebo
* Has a history of congestive heart failure (New York Heart Association [NYHA] Class 3 or 4)
* Has a history of myocardial infarction, uncontrolled arrhythmias, cardiac revascularization, unstable peripheral arterial disease and/or stroke within 6 months of screening
* History of significant multiple and/or severe allergies (e.g., food, drug, latex allergy), or has had an anaphylactic reaction or significant intolerability (i.e., systemic allergic reaction) to prescription or nonprescription drugs or food
* Has type 1 diabetes mellitus or secondary types of diabetes
* Has experienced complications of diabetes such as ketoacidosis, unstable diabetic retinopathy, or maculopathy
* Has previous or planned (during the trial period) obesity treatment with surgery or a weight loss device

Ages: 24 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-06-29 (Estimated); Study Completion 2026-06-29 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 42 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 28 days
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention.

SECONDARY OUTCOMES:
Plasma Concentration of MK-2828 at 24 Hours Postdose (C24) After Day 1 Dose | 24 hours post-Day 1 dose
  Blood samples will be collected to determine the C24 of MK-2828 in plasma after the Day 1 dose.
Plasma Concentration of MK-2828 at 24 Hours Postdose (C24) After Day 27 Dose | Predose on Day 28
  Blood samples will be collected to determine the C24 of MK-2828 in plasma after the Day 27 dose.
Change from Baseline in Placebo Corrected High-Sensitivity C-Reactive Protein (hsCRP) Serum Concentration | Baseline and Predose Day 28
  Blood samples will be collected to determine the change from baseline in placebo corrected hsCRP.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (11):
- United States (11):
  - ProSciento Inc. ( Site 0004), Chula Vista, California
  - California Clinical Trials Medical Group managed by PAREXEL ( Site 0008), Glendale, California
  - Velocity Clinical Research, Hallandale Beach ( Site 0010), Hallandale, Florida
  - Jacksonville Center for Clinical Research ( Site 0002), Jacksonville, Florida
  - Advanced Pharma CR, LLC ( Site 0001), Miami, Florida
  - QPS Miami Research Associates ( Site 0005), South Miami, Florida
  - AMR Lexington ( Site 0012), Lexington, Kentucky
  - Alliance for Multispecialty Research, LLC ( Site 0013), Kansas City, Missouri
  - Bio-Kinetic Clinical Applications, LLC dba QPS-MO ( Site 0009), Springfield, Missouri
  - AMR Clinical ( Site 0003), Knoxville, Tennessee
  - ICON Early Phase Services ( Site 0006), San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com